CLINICAL TRIAL: NCT03848637
Title: A Randomized, Open-label, Single Dose, 2-period, 2-treatment, Crossover Study to Compare the Pharmacokinetics and Safety/Tolerability of CKD-375 Tablet With D387 Tablet in Healthy Volunteers
Brief Title: The Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability of CKD-375
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 192BE18036
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): * Period 1: D387 (reference drug)
  * Period 2: CKD-387 (test drug)
  Interventions: Drug: CKD-375; Drug: D387
- Group 2 (Experimental): * Period 1: CKD-387 (test drug)
  * Period 2: D387 (reference drug)
  Interventions: Drug: CKD-375; Drug: D387

INTERVENTIONS:
Drug: CKD-375 — Test drug
Drug: D387 — Reference drug

SUMMARY:
The purpose of this clinical trial is to evaluate the pharmacokinetics and safety/tolerability after oral administration of CKD-375 and D387 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 to 55 years
2. Females who are not pregnant or breastfeeding or who have surgical infertility
3. Signed informed consent form
4. Other inclusion criteria, as defined in the protocol

Exclusion Criteria:

1. History of clinically significant hepatic, renal, nervous, immune, respiratory, endocrine, hemato-oncology, cardiovascular systemic disease or psychosis disorder
2. Clinical laboratory test values are outside the accepted normal range at Screening
3. Current smokers or those who cannot quit smoking during the period from 90 days before the first IP dosing to the last discharge.
4. Subject who drink excessive caffeine or alcohol continuously and who cannot discontinue caffeine or alcohol intake during the period from 3 days before the first IP dosing to the last discharge.
5. Participated in a clinical trial within 90 days prior to 1st IP dosing
6. Not eligible to participate for the study at the discretion of Investigator
7. Other exclusive inclusion criteria, as defined in the protocol

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-04-14 (Estimated); Primary Completion 2019-04-24 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration of Empagliflozin | Time Frame: 0 hour ~ 48 hour after drug administration
  Cmax of Empagliflozin
Maximum plasma concentration of Metformin | Time Frame: 0 hour ~ 48 hour after drug administration
  Cmax of Metformin
Area under the plasma concentration of Empagliflozin-time curve from time zero to time of last measurable concentration | Time Frame: 0 hour ~ 48 hour after drug administration
  AUClast of Empagliflozin
Area under the plasma concentration of Metformin-time curve from time zero to time of last measurable concentration | Time Frame: 0 hour ~ 48 hour after drug administration
  AUClast of Metformin

SECONDARY OUTCOMES:
Area under the plasma concentration of Empagliflozin-time curve from time zero to infinity | 0 hour ~ 48 hour after drug administration
  AUCinf of Empagliflozin
Area under the plasma concentration of Metformin-time curve from time zero to infinity | 0 hour ~ 48 hour after drug administration
  AUCinf of Metformin
Time to reach maximum (peak) plasma concentration of Empagliflozin following drug administration | 0 hour ~ 48 hour after drug administration
  Tmax of Empagliflozin
Time to reach maximum (peak) plasma concentration of Metformin following drug administration | 0 hour ~ 48 hour after drug administration
  Tmax of Metformin
Half-life of Empagliflozin | 0 hour ~ 48 hour after drug administration
  t1/2 of Empagliflozin
Half-life of Metformin | 0 hour ~ 48 hour after drug administration
  t1/2 of Metformin
Apparent clearance of Empagliflozin | 0 hour ~ 48 hour after drug administration
  CL/F of Empagliflozin
Apparent clearance of Metformin | 0 hour ~ 48 hour after drug administration
  CL/F of Metformin
Apparent volume of distribution of Empagliflozin | 0 hour ~ 48 hour after drug administration
  Vd/F of Empagliflozin
Apparent volume of distribution of Metformin | 0 hour ~ 48 hour after drug administration
  Vd/F of Metformin

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D, Principal Investigator — Seoul National University Hospital